CLINICAL TRIAL: NCT00716755
Title: The Minimal Effective Dose of Antipsychotic Medication in Older Patients With Schizophrenia: a PET Study.
Brief Title: Minimizing Doses of Antipsychotic Medication in Older Patients With Schizophrenia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Ariel Graff, MD, PhD, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156/2007
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Delusional Disorder; Psychotic Disorder
Keywords: Positron emission tomography; antipsychotics; risperidone; olanzapine; Dopamine; D2 receptor; elderly; schizophrenia; schizoaffective disorder; schizophreniform disorder; delusional disorder; psychotic disorder NOS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid; Mental Disorders | interventions — Risperidone; Olanzapine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Reduction (Experimental): See Intervention
  Interventions: Drug: Risperidone/Olanzapine and PET scans

INTERVENTIONS:
Drug: Risperidone/Olanzapine and PET scans — Current risperidone/olanzapine users who are 50 or older will be recruited. Dopamine D2 dopamine receptors using a selective D2 dopamine receptor ligand, [11C]-raclopride, and plasma levels of risperidone and 9-OH-risperidone, or of olanzapine, and prolactin will be measured on the 1st PET visit. Subsequently, there will be gradual dose reductions of risperidone or olanzapine by 0.5 and 2.5 mg per week, respectively (as long as the total reduction does not exceed 40%). At least 5 days after the termination of the dose taper, participants will have the second PET scan. Participants will be followed up for 24 weeks after the termination of the dose reduction.
  Other Names: Risperidal, Zyprexa

SUMMARY:
Since side effects of antipsychotics, dopamine D2 receptor blockers, frequently occur in older patients with schizophrenia and the risk is dose dependent, clinical guidelines universally advocate the use of lower doses. However, there is no report to test this dosing guideline with measurements of D2 receptor blockade caused by antipsychotics. In this study, dopamine D2 receptor occupancy will be measured, using Positron Emission Tomography (PET), in 40 patients aged 50 and older with schizophrenia-spectrum disorders before and after a gradual 40 % dose reduction of antipsychotics that was safely achieved in the past study while setting a target dose still above the lower limit of the dose range recommended in clinical guidelines for older patients. Our goal is to relate changes in clinical outcome, including subjective and objective clinical ratings, to dopamine D2 receptor occupancy, and compare these results with the data for younger patients in the literature.

DETAILED DESCRIPTION:
Antipsychotics play a central role in the treatment of schizophrenia irrespective of a patient's age. Aging is associated with an increased sensitivity to drug adverse effects, including adverse effects from antipsychotics. This concern is reflected in clinical guidelines recommending the use of lower doses of antipsychotics in elderly patients. For example, the Expert Consensus Guideline recommends dosing risperidone at 1.25 - 3.5 mg/d for older patients aged 65 and older with schizophrenia, compared with the recommended dose at 2.5 - 6.5 mg/d for younger patients. For olanzapine the recommended dose is 7.5 mg/day.

The risk for most adverse effects from antipsychotic drugs is dose-related and contributes to poor adherence and worse outcome. In addition to "objective" (in the sense of externally manifested) adverse effects including motor and autonomic side effects, it has been long been recognized that antipsychotics are also associated with a negative subjective sense of well-being that has been termed "neuroleptic dysphoria". This adverse effect has recently returned to the limelight in the literature since it has critical implications for adherence and recovery, and has also been associated with levels of striatal D2 receptor occupancy associated with motor side effects of both typical and atypical antipsychotics. Conceptually, therefore, it can be considered a subtle non-motor form of extrapyramidal symptoms (EPS) that may be manifested at doses lower than for motor EPS and may indeed represent the true "neuroleptic threshold" described by McEvoy two decades ago. Thus, optimal dosing of antipsychotic drugs (at clinical levels of D2 occupancy) would be expected to lead to better subjective experience, resulting in enhanced adherence to antipsychotic drugs.

Atypical antipsychotic drugs have been reported to show differential effects on weight gain and metabolic side effects, with an effect of dose established for olanzapine but not risperidone. The effect of dose on prolactin elevation has also been reported, which has raised concerns about the risk of osteoporosis and to a lesser extent breast carcinoma. Finally, motor side-effects are perhaps the best known dose-related consequence of antipsychotic drugs, and this is particularly true for risperidone. Lemmen et al. showed that higher doses of antipsychotics were reported to be associated with development to EPS in a combined analysis of 12 double-blind trials with risperidone, including 2,074 patients; moreover, the influence of this factor was more prominent in the elderly. Furthermore, higher cumulative amounts of prescribed antipsychotics have been reported to increase risks of developing tardive dyskinesia. These motor side-effects often not only impair the activities of daily living but also are expected to be associated with undesirable incidents such as falls and aspiration. In addition, EPS have been reported to be associated with cognitive dysfunction, although it is still uncertain of to what extent EPS affect this cognitive impairment directly and indirectly.

Risperidone and olanzapine are the most widely used antipsychotic drugs, and risperidone has been marketed for use of behavioral disturbance in dementia in the United States. Moreover, they are both available in generic form, making it more widely available. Our clinical experience, as well as preliminary data at CAMH, suggests that the dosing guidelines for elderly patients with schizophrenia may not be universally followed and patients' dosing may not necessarily be adjusted with age (personal communication, Dr Beth Sproule). Given the dose-related concerns, age-related sensitivity, and recent concerns about excess mortality in patients with dementia treated with atypical antipsychotics, it is both reasonable and standard practice to gradually reduce the dose of antipsychotics with increasing age in patients with schizophrenia. Gradual antipsychotic dose reduction was successfully completed in a naturalistic study, of carefully selected patients (n = 27) with schizophrenia and related psychotic disorders aged 45 years and older. A 40 % dose reduction (from mean dose 190 to 110 mg chlorpromazine equivalent) was tolerated by 70% of the sample who experienced no increase in psychotic symptoms after 6 months, suggesting that most older patients tolerate a lower dose of antipsychotic without adverse clinical outcome. Further, those subjects who demonstrated worsening of psychotic symptoms were stabilized within several days with a small increase in neuroleptic dosage over the last dosage on which the patient was stabilized and no patients required hospitalization. These results are consistent with the documented safety and clinical value of gradual antipsychotic dose reduction in younger patients with schizophrenia.

Previous PET studies in adult patients with schizophrenia have shown that clinical response is unlikely below striatal dopamine D2 receptor occupancy of 65 %, and conversely motor side effects very likely at occupancies in excess of 80 %. This therapeutic window for risperidone in terms of occupancy is consistent with the clinical therapeutic dose range of 2 - 6 mg, with the 2 mg dose barely reaching the occupancy threshold of 65 %. The lower dose range recommended by clinical guidelines for elderly patients with schizophrenia (1.25 - 3.5 mg for risperidone) suggests that the therapeutic window is lower for elderly patients. Thus dosing the antipsychotic at either the upper limits of this dose range, or above these limits would be expected to be associated with subjective or objective EPS, and warrants a trial of lower dosing as per guidelines. Indeed, Tort et al have simulated the relationship between plasma level and D2 occupancy for the atypical antipsychotic drugs based on their affinity for the D2 receptor and concluded that in the presence of EPS the antipsychotic dose could well be halved and the resultant D2 occupancy would be expected to stay well within the D2 occupancy therapeutic window of 65-80 %. If the elderly patients with schizophrenia do indeed respond and show maintenance of wellness at lower doses, this suggest one or more of the following mechanisms may be involved: (a) for a given dose they are reaching equivalent plasma levels as younger patients, (b) for a given plasma drug level they are achieving higher central occupancy, or (c) they show clinical response at a lower level of occupancy.

We propose a prospective study to assess dopamine D2 receptor occupancy before and after a gradual 40% dose reduction of risperidone and olanzapine that was safely achieve in patients over the age of 45 in a past study while setting a target dose above the lower limit of the dose range recommended in clinical guidelines, ie., 1.5 mg/day and 7.5 mg/day for risperidone and olanzapine respectively, for older patients. Our goal is to relate changes in clinical outcome, including subjective and objective clinical ratings, to striatal dopamine D2 receptor occupancy, and compare these results with the data for younger patients in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Age of 50 and older
* DSM-IV/SCID diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or psychotic disorder NOS
* Having been treated with oral risperidone at a steady dose of ≥ 2 mg/day, or with olanzapine at a steady dose of ≥10 mg/day, for at least 12 months.

Exclusion Criteria:

* Incapacity to provide consent to psychiatric treatment
* Participation in this study would result in exceeding the annual radiation dose limits (20 mSv) for human subjects participating in research studies.
* Substance abuse or dependence (within past six months)
* Positive urine drug screen
* Positive serum pregnancy test at screening or positive urine pregnancy test before PET scan
* Having taken more than one dose of antipsychotics other than risperidone or olanzapine during the 7 days preceding the PET scan
* History of treatment with long-acting (depot) neuroleptic antipsychotic medication or Risperdal Consta within 12 months of PET scanning
* Metal implants or a pace-maker that would preclude the MRI scan
* Addition of or change in dose of antidepressants, valproic acid, lithium, carbamazepine, or lamotrigine for mental health reasons within 12 months of screening
* History of head trauma resulting in loss of consciousness > 30 minutes that required medical attention
* Unstable physical illness or significant neurological disorder including a seizure disorder
* Size of head, neck, and body being unable to fit PET and MRI scanners
* Refusal to give consent to investigator to communicate with physician of record for the entire duration of the study
* Psychiatric concerns raised by the physician of record regarding participation in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Occupancy of risperidone/olanzapine at the dopamine D2 receptor | intermittently
  PET scan data showing how much dopamine D2 receptors are occupied

SECONDARY OUTCOMES:
Tolerability of 40 % antipsychotic dose reduction and its relation to the % change in occupancy following dose reduction | intermittent
  Clinical assessment data on how well the antipsychotic dose reduction is tolerated and its relationship to the PET scan data
Relationship between plasma concentration of risperidone and its active metabolite, 9-OH-risperidone(or olanzapine) and dopamine D2 receptor occupancy in older patients, in comparison to historic young controls. | intermittent
  Antipsychotic levels in the blood and its relationship to the PET scan data and to healthy control data

CONTACTS AND LOCATIONS:
Overall Officials: David C. Mamo, MD MSc, Principal Investigator — Centre for Addiction and Mental Health; Ariel Graff-Guerrero, MD,PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iwata Y, Nakajima S, Caravaggio F, Suzuki T, Uchida H, Plitman E, Chung JK, Mar W, Gerretsen P, Pollock BG, Mulsant BH, Rajji TK, Mamo DC, Graff-Guerrero A. Threshold of Dopamine D2/3 Receptor Occupancy for Hyperprolactinemia in Older Patients With Schizophrenia. J Clin Psychiatry. 2016 Dec;77(12):e1557-e1563. doi: 10.4088/JCP.15m10538. PMID 28086010
- [Derived] Fervaha G, Caravaggio F, Mamo DC, Mulsant BH, Pollock BG, Nakajima S, Gerretsen P, Rajji TK, Mar W, Iwata Y, Plitman E, Chung JK, Remington G, Graff-Guerrero A. Lack of association between dopaminergic antagonism and negative symptoms in schizophrenia: a positron emission tomography dopamine D2/3 receptor occupancy study. Psychopharmacology (Berl). 2016 Oct;233(21-22):3803-3813. doi: 10.1007/s00213-016-4415-6. Epub 2016 Aug 24. PMID 27557949
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre. — http://www.camh.net/research